CLINICAL TRIAL: NCT03424278
Title: Efficacy of Motor Control Exercises and Resistance Training on Pain, Function, Kinesiophobia and Trunk Strength in Individuals With Non-specific Chronic Low Back Pain
Brief Title: Efficacy of Exercises in Individuals With Non-specific Chronic Low Back Pain
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The participants recruitment was to difficult
Sponsor: University of Brasilia (Other)
Collaborators: Military Fire Department of the Federal District (Unknown)
Responsible Party: Principal Investigator, Wagner Rodrigues Martins, Professor, University of Brasilia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PPGCR1
Record Dates: First submitted 2018-01-31; First posted 2018-02-06 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2021-01

CONDITIONS: Low Back Pain
Keywords: Low back pain; Exercise
MeSH Terms: conditions — Low Back Pain; Motor Activity

STUDY DESIGN:
Intervention Model Description: Parallel randomized controlled trial.
Who Masked: Outcomes Assessor
Masking Description: An assessor who don't now in which groups the participants has been allocated.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motor Control (Active Comparator)
  Interventions: Other: Motor control exercises
- Resistance Training (Experimental)
  Interventions: Other: Resistance training exercises

INTERVENTIONS:
Other: Motor control exercises — Motor control exercises for the deep trunk muscles in patients with chronic low back pain is based on evidence of motor control dysfunction, including delayed onset of activity in the transversus abdomens and internal oblique abdominal muscles and segmental hypertrophy of the lumbar multifidus muscle.
  Arms: Motor Control
Other: Resistance training exercises — A type of strength-building exercise program that requires the body muscle to exert a force against some form of resistance, such as weight, stretch bands, water, or immovable objects. Resistance exercise is a combination of static and dynamic contractions involving shortening and lengthening of skeletal muscles.
  Arms: Resistance Training

SUMMARY:
This is a randomized controlled trial project to analyze the effectiveness of lumbar motor control exercises and lumbar resistance training on pain, functional, kinesiophobia and trunk strength in individual with chronic low back pain. The project has two parallel arms and will be supervised by physiotherapists (motor control exercises) and physical education professionals (resistance training). The participants will be Militaries of the Military Fire Department of the Federal District who presents in the recruitment regular low back pain more than 3 months. The two groups will be supervised in12 weeks of exercises in the Physical Activity Center of Military Fire Department of the Federal District. Our hypotheses is that the resistance training effects wil be superior to motor control exercises only for trunk strength (isokinetic flexion and extension).

ELIGIBILITY:
Inclusion Criteria:

* Nonspecific chronic low back pain (defined as pain and discomfort) localized below the costal margin and above the inferior gluteal folds, with or without referred leg pain of at least 3 months' duration.

Exclusion Criteria:

* Spinal pathology (eg, tumor, infection, fracture, inflammatory disease), pregnancy, nerve root compromise, previous spinal surgery, major surgery scheduled during treatment or follow-up period, and presence of any contraindication to exercise.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2017-02-10 (Actual); Primary Completion 2017-02-10 (Actual); Study Completion 2017-11-10 (Estimated)

PRIMARY OUTCOMES:
Numerical Rating Scale (NRS) | One day
  In a Numerical Rating Scale (NRS), patients are asked to circle the number between 0 and 10, 0 and 20 or 0 and 100 that fits best to their pain intensity. Zero usually represents 'no pain at all' whereas the upper limit represents 'the worst pain ever possible'.
Roland-Morris Disability Questionnaire (RDQ) | One day
  Questionnaires to measure and monitor changes in functional outcome in patients with LBP. The RDQ evaluates 24 activity limitations due to LBP, while the ODI consists of 10 items assessing the level of pain interference with physical activities.
Tampa Scale for Kinesiophobia (TSK) | One day
  Measures the excessive, irrational, and debilitating fear of movement and activity resulting from a feeling of vulnerability to painful injury or re-injury. Its a 17-item scale.

SECONDARY OUTCOMES:
Trunk Muscle strength | One day
  This outcome will be assessed by a isokinetic dynamometer. Today dynamometry routinely assesses muscle performance in healthy and symptomatic populations.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Brasilia, Brasília, Federal District, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Saragiotto BT, Maher CG, Yamato TP, Costa LOP, Costa LCM, Ostelo RWJG, Macedo LG. Motor Control Exercise for Nonspecific Low Back Pain: A Cochrane Review. Spine (Phila Pa 1976). 2016 Aug 15;41(16):1284-1295. doi: 10.1097/BRS.0000000000001645. PMID 27128390
- [Background] Saragiotto BT, Maher CG, Yamato TP, Costa LO, Menezes Costa LC, Ostelo RW, Macedo LG. Motor control exercise for chronic non-specific low-back pain. Cochrane Database Syst Rev. 2016 Jan 8;2016(1):CD012004. doi: 10.1002/14651858.CD012004. PMID 26742533
- [Background] Bystrom MG, Rasmussen-Barr E, Grooten WJ. Motor control exercises reduces pain and disability in chronic and recurrent low back pain: a meta-analysis. Spine (Phila Pa 1976). 2013 Mar 15;38(6):E350-8. doi: 10.1097/BRS.0b013e31828435fb. PMID 23492976
- [Background] Chang WD, Lin HY, Lai PT. Core strength training for patients with chronic low back pain. J Phys Ther Sci. 2015 Mar;27(3):619-22. doi: 10.1589/jpts.27.619. Epub 2015 Mar 31. PMID 25931693
- [Background] Steele J, Bruce-Low S, Smith D. A review of the clinical value of isolated lumbar extension resistance training for chronic low back pain. PM R. 2015 Feb;7(2):169-87. doi: 10.1016/j.pmrj.2014.10.009. Epub 2014 Oct 29. PMID 25452128
- [Background] Kristensen J, Franklyn-Miller A. Resistance training in musculoskeletal rehabilitation: a systematic review. Br J Sports Med. 2012 Aug;46(10):719-26. doi: 10.1136/bjsm.2010.079376. Epub 2011 Jul 26. PMID 21791457